CLINICAL TRIAL: NCT06612697
Title: Long-Term Outcomes of Early-Stage Nasopharyngeal Carcinoma Patients Treated with Radiotherapy Alone
Status: Active, not recruiting | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE23408A
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Nasopharyngeal Carcinoma (NPC); Oncology; Radiology
Keywords: nasopharyngeal carcinoma; early-stage; Radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Neoplasms | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Radiology — A retrospective analysis was conducted using systematic records from the Department of Radiation Oncology at our hospital. The study included patients diagnosed with nasopharyngeal carcinoma through endoscopic pathological reports from January 1, 1984, to December 31, 2022. Eligible patients had baseline imaging (CT or MRI) prior to treatment, received definitive radiotherapy at our institution, and were followed up long-term with complete medical records.

SUMMARY:
Nasopharyngeal carcinoma (NPC) is a malignant tumor primarily originating in the nasopharynx, commonly found in populations in southern China, certain regions of Asia, and North Africa. The main treatment for NPC is primarily radiotherapy, with some patients receiving combined chemotherapy. Early-stage NPC patients can achieve adequate tumor control with radiation therapy alone. Various studies report that the 5-year survival rate for very early-stage NPC exceeds 90%. However, some stage I patients experience local recurrence or distant metastasis after treatment, indicating treatment failure. This study aims to retrospectively analyze the factors contributing to treatment failure and prognostic factors in this group of early-stage NPC patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with nasopharyngeal carcinoma based on endoscopic pathological reports.
* Included early-stage patients classified as cT1-2, cN0-1, M0.
* Had baseline imaging (CT or MRI) prior to treatment.
* Received definitive radiotherapy at our institution and had long-term follow-up with complete medical records.

Exclusion Criteria:

* Excluded from the study are patients with local lymph node metastasis or distant metastasis (cN ≥ 2, M = 1) as determined by imaging studies.
* Patients who did not receive definitive radiotherapy at our institution or had incomplete medical records during long-term follow-up are also excluded.
* Patients diagnosed with any other primary cancer within five years prior to the diagnosis of nasopharyngeal carcinoma (excluding DCIS and skin cancer) are excluded from the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective analysis was conducted on patients diagnosed with nasopharyngeal carcinoma based on endoscopic pathological reports at our institution from January 1, 1984, to December 31, 2022. Eligible patients had baseline imaging (CT or MRI) prior to treatment, received definitive radiotherapy at our institution, and had long-term follow-up with complete medical records.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | The 5-year survival rate after surgery
  Overall survival is an important indicator for assessing treatment efficacy, reflecting the impact of treatment on extending patient life. It is typically calculated by measuring the time from the start of treatment until the patient's death or loss to follow-up.
Disease-Free Survival | Within 5 years after surgery
  Disease-free survival (DFS) refers to the period during which a patient remains free of disease recurrence following treatment. This indicator helps evaluate the effectiveness of the treatment, particularly in early-stage cancer patients, as it reflects the durability of tumor control. DFS is typically calculated by measuring the time from the end of treatment to the first occurrence of disease recurrence.
Local Control Rate | Within 5 years after surgery
  Local control rate refers to the effectiveness of treatment in managing the tumor at its primary site, reflecting the ability to prevent local recurrence. A high local control rate indicates that the treatment has successfully eradicated the tumor or effectively suppressed its growth, which is crucial for the prognosis of tumors such as nasopharyngeal carcinoma.

SECONDARY OUTCOMES:
Recurrence Rate | Within 5 years after surgery
  Recurrence rate refers to the proportion of patients who experience tumor recurrence after treatment, encompassing both local recurrence and distant metastasis. This indicator aids in evaluating the overall effectiveness of the treatment and identifying potential prognostic factors, while also revealing differences between various treatment methods.
Metastasis Rate | Within 5 years after surgery
  Metastasis rate refers to the proportion of tumors that spread to other sites in the body. This indicator provides information about disease progression. A high metastasis rate may suggest more aggressive biological characteristics of the tumor and can influence the choice of treatment strategies.
Treatment-Related Adverse Events | Within 5 years after surgery
  Treatment-related adverse events refer to the side effects or complications that patients experience during the course of treatment. These events can affect the patient's quality of life and the continuity of treatment, making it crucial to understand their incidence and nature in order to assess the overall safety of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan